CLINICAL TRIAL: NCT02217449
Title: Virtual Chromoendoscopy for Distal Polyps
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0010
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- HD: Prediction of histology
  Interventions: Other: Prediction of histology
- Virtual Chromoendoscopy: Prediction of histology
  Interventions: Other: Prediction of histology

INTERVENTIONS:
Other: Prediction of histology

SUMMARY:
To assess the accuracy of predicting histology with virtual chromoendoscopy for distal colorectal polyps according to the ASGE PIVI statement.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Screening or surveillance colonoscopy

Exclusion Criteria:

* history of inflammatory bowel disease
* poor bowel preparation
* colectomy
* anticoagulation
* polyposis syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing screeining or surveillance colonoscopy
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Effectivity of virtual chromoendoscopy | 3 years
  Upon visualization of a polyp in white-light, the location and size (as compared to open biopsy forceps or snare) are noted. Afterwards, virtual chromoendoscopy is used to visualize and enhance the mucosal vascular pattern and the mucosal surface pattern morphology of the polyp. The endoscopist makes a real time assessment of each polyp according to size, shape, Paris classification and surface characteristics including pit pattern and mucosal vascular pattern morphology, colour, and type of depression. Further, the endoscopist is assigning a level of confidence (high or low) to each real time prediction. Afterwards, all polyps are resected using standard techniques and processed for pathological evaluation. Each polyp is assessed by an experienced GI pathologist blinded to the real time prediction of polyp histology. Finally, real time and histological results are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Rath T, Tontini GE, Nagel A, Vieth M, Zopf S, Gunther C, Hoffman A, Neurath MF, Neumann H. High-definition endoscopy with digital chromoendoscopy for histologic prediction of distal colorectal polyps. BMC Gastroenterol. 2015 Oct 22;15:145. doi: 10.1186/s12876-015-0374-3. PMID 26493200